CLINICAL TRIAL: NCT03977649
Title: A RandomizEd, Double-blind, Cross-over Study to Assess Erenumab effecT on BRAIN Networks Function and Structure in Comparison to Placebo in Episodic Migraine Patients
Brief Title: A Functional MRI Study on Erenumab Treatment Effects in Episodic Migraine Patients
Acronym: RESET BRAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAMG334AIT03
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Migraine Disorders
Keywords: AMG334; erenumab; functional MRI; connectivity
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Intervention Model Description: After a run-in phase of 4 weeks, patients will be randomized, according to a 1:1 ratio, to a 24 weeks of treatment, as follow:
  * Sequence 1: A/B
  * Sequence 2: B/A where: A=monthly subcutaneous erenumab 140 mg for 12 weeks; B=monthly subcutaneous masked placebo for 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study treatments will be all identical in packaging, labeling, schedule of administration, appearance, taste and odor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- erenumab (Experimental): monthly subcutaneous erenumab 140 mg for 12 weeks
  Interventions: Drug: erenumab
- placebo (Placebo Comparator): monthly subcutaneous masked placebo for 12 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: erenumab — erenumab 140 mg sc every 4 weeks
  Arms: erenumab
Drug: placebo — placebo sc every 4 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the effects of erenumab on central sensitization and brain networks connectivity of migraine patients

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo-controlled trial with a 2-sequence, 2-period, 2-treatment crossover design. The study population will consist of adult male and female subjects with a documented history of episodic migraine (4 to 14 baseline migraine days), who have failed at least 2 previous migraine prophylactic treatment for lack of efficacy or tolerability. After a run-in phase of 4 weeks, patients will be randomized, according to a 1:1 ratio, to a 24 weeks of treatment, as follow:

* Sequence 1: A/B
* Sequence 2: B/A where: A=monthly subcutaneous erenumab 140 mg for 12 weeks; B=monthly subcutaneous masked placebo for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study History of migraine with or without aura for at least 12 months prior to screening 4. Migraine frequency: ≥ 4 and < 15 migraine days per month on average across the 3 months prior to screening and confirmed during the baseline phase based on diary calculation
* Headache frequency: <15 headache days per month on average across the 3 months prior to screening and confirmed during the baseline phase based on diary calculation
* Failure to 2 or more previous treatment categories locally indicated for migraine prophylaxis due to either lack of efficacy or poor tolerability

Exclusion Criteria:

* History of cluster headache or hemiplegic migraine headache
* History of chronic pain disorders and neuropathic pain
* History of head trauma or seizure or major psychiatric disorders or suicidal ideation/behavior at any time before screening
* Currently, receiving any other prophylactic treatment for migraine and/or prohibited medications, non-pharmacologic interventions or devices (any substance, non-pharmacologic intervention or device acting at central nervous system), or less than 60 days or 5 half-lives prior to the start of the baseline period, during the baseline period, or treatment period
* Exposure to botulinum toxin in the head and/or neck region within 4 months prior to the start of the baseline period, during the baseline period, or treatment period.
* Taken the following for any indication in any month during the 2 months prior to the start of the baseline period:

  * Ergotamines or triptans on ≥ 10 days per month, or
  * Simple analgesics (non-steroidal anti-inflammatory drugs [NSAIDs], acetaminophen) on ≥ 15 days per month, or
  * Opioid- or butalbital-containing analgesics on ≥4 days per month.
* Previous exposure to erenumab or exposure to any other prophylactic CGRP-targeted therapy (prior to and during the study)
* History or evidence of any other unstable or clinically significant medical condition that in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
* Subject has any clinically significant vital sign, laboratory, or electrocardiogram (ECG) abnormality during screening that, in the opinion of the investigator, could pose a risk to subject safety or interfere with the study evaluation
* Evidence of drug or alcohol abuse or dependence within 12 months prior to screening, based on medical records or patient self-report
* Pregnant or breastfeeding
* All the clinical conditions for which undergoing an MRI scan is contraindicated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
z-score maps change difference between-treatment-groups | baseline, month 3, month 6
  z score maps are measures of resting state functional connectivity strength in the brain areas involved in pain processing
z-score maps difference between clinical response groups within the two treatment groups. | baseline, month 3, month 6
  clinical response assessed as reduction by 50% in monthly migraine days ,MMD, in the last month vs baseline.
  z score maps relative to resting state functional connectivity strength in the brain areas involved in pain processing

SECONDARY OUTCOMES:
Correlation (by treatment groups and in all patients) between the changes in the resting state functional connectivity strength, measured as z-score maps, and clinical outcomes | month 3, month 6
  clinical outcomes: the percentage of change in monthly migraine, b. the reduction in monthly average severity of migraine pain, c. the percentage of reduction in monthly number of days with use of acute treatments, d. the change in HIT-6 score
Between-treatment-groups difference in change of resting state functional connectivity strength, from baseline to month 3 of treatment, measured as z-score maps. in the brain regions involved in migraine symptoms | baseline, month 3, month 6
  migraine symptoms: a. sensory hypersensitivity (allodynia) b. visual or auditory hypersensitivity (photophobia or phonophobia) c. neurovegetative symptoms (nausea) d. altered emotional control of pain
Correlation (by treatment group and in all patients) between of the changes in the resting state functional connectivity strength of the areas involved in migraine symptoms and the reduction of the respective symptoms | month 3, month 6
  the clinical response here is described as reduction of the migraine symptoms: changes in the Allodynia Symptom Checklist 12 (ASC-12) score as measure of allodynia, the percentage changes in number of days with photophobia and phonophobia, and the percentage changes in number of days with nausea, changes in HADS score as measure of anxiety and depressive behaviour
Baseline resting state functional connectivity strength will be evaluated by treatment group and in all patients as potential predictors of treatment clinical response defined by the achievement of at least 50% reduction of monthly migraine days | baseline, month 3, month 6
  baseline functional MRI markers predictive of good clinical response to erenumab
Changes in z-score maps from baseline to month 3 of erenumab treatment and from baseline to month 6 with 3 months with erenumab followed by 3 months of placebo | baseline, month 3, month 6
  the effects of the erenumab discontinuation on fMRI after 3 months of placebo treatment

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, L’Aquila
  - Novartis Investigative Site, Napoli

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com